CLINICAL TRIAL: NCT01703156
Title: Stress Testing Versus Non-Stress Testing Based Strategy in Patients Hospitalized With Low-Risk Acute Coronary Syndromes: A Randomized, Single-Center Pilot Study
Brief Title: Low Risk Acute Coronary Syndrome
Acronym: LOW ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mazen Abu-Fadel, M.D., Associate Professor of Medicine, University of Oklahoma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Low Risk ACS; IRB#14542 (Other: University of Oklahoma Health Sciences Center Institutional Review Board)
Record Dates: First submitted 2012-10-03; First posted 2012-10-10 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Low Risk Acute Coronary Syndrome
Keywords: Low Risk ACS, Acute Coronary Syndrome, Stress Testing, Non-Stress Testing
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-Stress Group (Experimental): Medical therapy will be implemented and will include the following: aspirin, clopidogrel, b-blockers, and statins. The dosages of aspirin, b-blocker and statin will be left to the discretion of the treating physician. Statins will be initiated irrespective of LDL unless contraindicated. Clopidogrel will be taken for at least one month and ideally up to one year. Sublingual nitroglycerin will be provided to all patients. Other anti-ischemic medications including long-acting nitrates, calcium channel blockers, and ranolazine may be provided at the treating physicians' discretion. If a patient has contraindications to any medications, they will not be administered. If a statin contraindication exists, other cholesterol-lowering medications may be administered. Appendix 4 shows the detailed management of low risk ACS patients randomized to the non-stress group.
  Interventions: Procedure: No Stress Test
- Stress Group (Active Comparator): Medical therapy will be implemented and will include the following: aspirin, clopidogrel, b-blockers, and statins. Statins will be initiated irrespective of LDL unless contraindicated. Clopidogrel will be taken for at least one month and ideally up to one year. Sublingual nitroglycerin will be provided to all patients. Other anti-ischemic medications including long-acting nitrates, calcium channel blockers, and ranolazine may be provided at the treating physicians' discretion. If a statin contraindication exists, other cholesterol-lowering medications may be administered. All patients will undergo noninvasive stress testing. Results of individual stress tests will be reviewed by a cardiologist. Based on the myocardium deemed at risk and patient symptoms, further testing with angiography and revascularization using percutaneous techniques and/or coronary artery bypass grafting may be considered. Likewise, medical treatment may be adjusted.
  Interventions: Procedure: Stress Test

INTERVENTIONS:
Procedure: Stress Test
  Arms: Stress Group
Procedure: No Stress Test
  Arms: Non-Stress Group

SUMMARY:
A large number of patients are diagnosed with low risk ACS, and these individuals are at significant cardiovascular risk. Though guidelines recommend stress testing to manage low risk ACS patients, evidence supporting this recommendation is not based on trials examining this population. A well-designed, randomized trial is warranted to determine if stress testing is useful in managing low risk ACS. If medical therapy alone is equivalent as the investigators hypothesize, healthcare expenditures could be reduced and patients may not be exposed to the harms associated with more invasive cardiac testing such as coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

1. TIMI score < or = to 2(12)
2. TIMI risk score of 3 with no known CAD, greater than 50% in one or more vessels
3. Normal cardiac biomarkers (3 sets over 12-88 hours)
4. No evidence of acute ischemia on electrocardiograms
5. Normal ejection fraction (>40%) on echocardiography
6. Age 30-75
7. Ability to complete noninvasive stress test
8. Ability to provide informed consent

Exclusion Criteria:

1. Presence of another medical condition to explain chest pain or non-cardiac chest pain (i.e. pneumonia, costochondritis)
2. Any patient who is initially classified as low risk but whom develops recurrent symptoms of ischemia, hemodynamic instability, or arrhythmias attributable to ischemia
3. Evidence of ischemia on electrocardiogram
4. Abnormal cardiac biomarkers
5. History of medical noncompliance or social circumstances preventing compliance
6. Life span estimated at <1 year
7. Pregnancy
8. Refusal to sign consent

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality, hospitalization for UA/NSTEMI or STEMI, and urgent revascularization | one year
  Primary endpoints include the composite of all-cause mortality, hospitalization for Unstable Angina/Non ST-Elevation Myocardial Infarction (UA/NSTEMI) or ST-Elevation Myocardial Infarction (STEMI), and urgent revascularization (coronary artery bypass grafting or percutaneous coronary intervention).

SECONDARY OUTCOMES:
Secondary endpoints will include mortality, UA/NSTEMI or STEMI, coronary revascularization, unplanned diagnostic coronary angiography, noninvasive stress testing, medication adjustments, and medication side effects. | one year
  Secondary endpoints will include: mortality, UA/NSTEMI or STEMI, coronary revascularization, unplanned diagnostic coronary angiography, noninvasive stress testing, medication adjustments, and medication side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen S Abu-Fadel, MD, FACC, FSCAI, Principal Investigator — OUHSC and VAMC OKC
Locations (1):
- Veteran's Affairs Medical Center, Oklahoma City, Oklahoma, United States